CLINICAL TRIAL: NCT04139447
Title: Analysis of the Distribution of Adrenal Steroids in Blood and Urine Measured by Mass Spectrometry Coupled to Liquid Chromatography in a Control Population
Brief Title: DAnalysis of the Distribution of Adrenal Steroids in a Control Population
Acronym: STEROTEM
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: AREM (Association Régionale Endocrinologie Métabolisme) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2013_11; 2013-A01632-43 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2019-01-14; First posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Adrenal Disease
Keywords: Adrenal steroids; mass spectroscopy; liquid chromatography
MeSH Terms: conditions — Adrenal Gland Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum, urine.
  * blood ionogram, serum creatinine, CO2T (heparin tube)
  * Plasma Renin Activity 5PRA)
  * Steroid blood (B, 18-OH B, DOC, 18-OH DOC, S, F, 18-OH F, 17-OH progesterone, 21-deoxycortisol, delta 4 androstenedione, 17-OH pregnenolone, aldosterone, SDHA)
  * Urine ionogram (natriuresis, kaliuresis)
  * Steroid Urine (E, F, THF, aTHF, THE, aldosterone)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy subjects

SUMMARY:
This is a biomedical research study on the determination of adrenal steroids. It has been proposed in recent years as a tool for the diagnostic orientation of an adrenal pathology. The main objective is to analyze the distribution of blood and urinary adrenal steroid values in a population of 60 controls. The secondary objective is to establish reference values for each of these parameters, if their distribution permits, and to study the possible link between the blood pressure level, the orthostatism state, the potassium level and these adrenal steroids.

ELIGIBILITY:
Inclusion Criteria:

* Negative blood pregnancy test
* Normosalt diet
* Men and women ≥ 18 years
* Being able and willing to give written informed consent

Exclusion Criteria:

* Personal history of diabetes, high blood pressure, adrenal pathologies.
* Family history of adrenal pathologies.
* Taking of the following drugs:

Antihypertensives drugs: ACE inhibitor, Angiotensin II receptor, beta-blocker, thiazide diuretic, loop diuretic, anti-aldosterone, dihydropyridine-type calcium antagonist.

* Hormone replacement therapy, cyproterone acetate
* NSAID (except occasional intake), corticosteroid
* Antidepressant: serotonin reuptake inhibitor (paroxetine, fluoxetine, sertraline, citalopram)
* Contraception or estrogen / progestin treatment (progestins only allowed)
* Not be able to keep standing position.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Biomedical research to analyze the distribution of blood and urinary adrenal steroid values in a population of 60 healthy controls.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
difference of the distribution of blood steroid values in a population control group | At baseline
  The value will be measured by mass spectrometry coupled with liquid chromatography (HPLC-MS) and 16 global parameters will be analyses (B, 18-OH B, DOC, 18-OH DOC, S, F, 18-OH F, 17-OH progesterone, 21-desoxycortisol, delta 4 androstenedione, 17OHpregnenolone, aldosterone, SDHA, E, testosterone, estradiol
difference of the distribution of urinary steroid values in a population control group | At baseline
  The value will be measured by mass spectrometry coupled with liquid chromatography (HPLC-MS) and 6 global parameters will be analyses (E, F, THF, aTHF, THE, aldosterone)

SECONDARY OUTCOMES:
Blood pressure taken while sitting, lying or standing | At baseline
blood concentration of kaliemia | at baseline

CONTACTS AND LOCATIONS:
Overall Officials: Claire Douillard, MD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU, Hôpital Claude Huriez, Lille, France